CLINICAL TRIAL: NCT03186534
Title: Efficacy of Couples-Based HIV Prevention in Vulnerable Young Men
Brief Title: Randomized Trial of an HIV Prevention and Relationship Education Program for Young Male Couples
Acronym: 2GETHER
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: University of Cincinnati (Other); Howard Brown Health Center (Other)
Responsible Party: Principal Investigator, Michael E. Newcomb, Assistant Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: R01AA024065 (NIH)
Record Dates: First submitted 2017-06-12; First posted 2017-06-14 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Hiv; Chlamydia; Gonorrhea; Relation, Interpersonal
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Chlamydia Infections; Gonorrhea

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 2GETHER (Experimental): 2GETHER is an HIV prevention and relationship education program designed for young male couples. 2GETHER consists of 4 sessions (2 group sessions, 2 individualized couple session) administered over the course of 1 month (1 session per week). Group sessions focus on developing skills related to sexual health and relationship functioning, including HIV prevention in couples, communication skills, coping skills, problem-solving and acceptance. Individualized couple sessions focus on implementation of skills specific to the needs of each couple.
  Interventions: Behavioral: 2GETHER
- Positive Affect Enhancement (Active Comparator): The control condition is a positive affect enhancement program for couples. This is an active and attention-matched control condition. Group sessions focus on developing various coping skills that aim to enhance positive emotions in couples, and individualized couple sessions focus on skills implementation.
  Interventions: Behavioral: Positive Affect Enhancement

INTERVENTIONS:
Behavioral: 2GETHER — Communication skills, coping skills, problem-solving, acceptance, HIV prevention
  Arms: 2GETHER
Behavioral: Positive Affect Enhancement — coping skills for enhancing positive emotions, mindfulness
  Arms: Positive Affect Enhancement

SUMMARY:
Young gay, bisexual, and other men who have sex with men (YMSM) are the only risk group in which rates of new HIV infections are on the rise. There has been a relative dearth of research dedicated to understanding these health disparities between gay/bisexual and heterosexual youth, and even less has focused on identifying factors that might promote resilience against negative health outcomes. Understanding both risk factors and processes of resilience is critical in developing efficacious interventions to improve health in this population.

Through a grant from the National Institutes of Health, the investigators completed formative research with young male couples. Qualitative interviews identified preferences for couples-based intervention format and content. While coupled YMSM expressed some interest in HIV prevention, participants were most interested in building relationship skills. Coupled YMSM preferred group-based interventions in order to meet and learn from other couples but had concerns about discussing personal topics in groups. Quantitative analyses found that the rate of condomless sex in couples increased from adolescence to young adulthood. Further, the influence of older partners, partner violence, and drinking before sex were strongest in emerging adulthood. Informed by these, the research team developed 2GETHER, which aims to reduce HIV transmission risk in couples by enhancing relationship functioning. 2GETHER is a four session program. The first two sessions are group sessions aimed at skills building, and the second two sessions are individualized couple sessions aimed at skills implementation. Modules address communication skills, coping with stress (both general and sexual minority-specific stress), relationship sexual satisfaction, and HIV transmission risk within the dyad and with outside partners. 2GETHER was designed to address HIV transmission risk in couples regardless of HIV status; couples learn to use behavioral and biomedical approaches to prevent both HIV acquisition (e.g., HIV testing, condom use, pre-exposure prophylaxis) and transmission (e.g., medication adherence to reduce viral load), with an overarching emphasis on the health of the couple.

The investigators completed a pilot trial of 2GETHER with funding from Northwestern University. The pilot trial enrolled 57 couples (N=114) and demonstrated feasibility, acceptability, and preliminary efficacy of 2GETHER. This pilot trial used a non-randomized pre-/post-test design because the goal was to evaluate feasibility, acceptability and preliminary effects in a large number of diverse couples to inform a future efficacy RCT. Post-test occurred 2 weeks post-intervention, or ~2 months post-baseline. The pilot trial recruited a diverse sample of couples in less than one year and each program module receive high ratings of acceptability during post-sessions evaluation and an exit interview. At the 2-week post-test, the investigators observed significant decreases in HIV risk behavior, improvements in motivation to reduce HIV risk, and improvements in relationship investment.

The current study will conduct a randomized controlled trial (RCT) to test the efficacy of 2GETHER, a novel couples-based intervention for young men who have sex with men (YMSM) that aims to reduce HIV transmission risk by optimizing relationship functioning. The investigators will conduct an RCT with 200 dyads (total individual N=400), who will be randomized to receive the 2GETHER intervention or an attention-matched couples-based positive affect promotion program.

DETAILED DESCRIPTION:
The investigators will conduct a randomized controlled trial (RCT) with 200 dyads (total individual N=400), who will be randomized to receive the 2GETHER HIV prevention and relationship education intervention or an attention-matched couples-based positive affect enhancement program. Each program (both 2GETHER and control) delivers 4 sessions over 1-month; 2 group sessions of 4-8 couples focused on relationship skills building, and 2 individual couple sessions focused on skill utilization. Couples complete skills practice homework between sessions and receive community-based resources.

Eligibility Screening. Participants will be screened either online, over the phone with a member of the study staff, or in-person at Howard Brown Health Center, depending on the mode of recruitment (recruitment activities described below). (a) Online screening - young men who have sex with men (YMSM) who are recruited via social media ads or via email contact (i.e., email listservs, HBHC Primary Care patients) will be linked directly to the online eligibility screener, and YMSM recruited from flyer postings will be given a URL and the option to screen online. Potential participants will be greeted with a brief description of the project and will be asked if they are willing to answer some questions to assess their eligibility. Those who agree to participate will answer questions about their age, gender, and relationship status. Participants who meet initial eligibility criteria will be shown a message telling them that they are preliminarily eligible for the study. These participants will be asked to provide contact information for themselves and for their partner. If they do not consent to give contact information for their partner, the participant will be responsible for ensuring the partner also completes the screener. If they provide contact information for their partner, study staff will contact the partner and provide him with a link to complete the screener. (b) Phone screening - YMSM who opt to call the study phone number on the flyer will be screened by a study staff member. They will be given an overview of the study, the ability to ask questions, and will then be asked if they are interested in participating and asking their partner to participate. If they agree, the staff member will administer the online screener over the phone. All other procedures are analogous to the online screening. (c) In-person screening at Howard Brown Health Center - Upon completion of their HIV testing and counseling session or their primary care visit at Howard Brown, YMSM will be provided with a brief description of the 2GETHER project asked if they are interested in participating in the study. If interested, participants will complete the online eligibility screener. All other eligibility screener procedures are analogous to those described above for online screening. Screening data will be retained during the course of the study in order to help identify duplicate participants or participants faking eligibility.

Couple Confirmation. In order to participate in this study, both partners in the couple must complete the screener, meet all eligibility criteria, and be confirmed by study staff to be an actual couple. Couple confirmation will involve separate calls to each partner with a series of questions to elicit information about the individual, his partner, and their relationship (i.e., information only an actual couple would know about one another). After these phone calls, study staff will review the responses to determine agreement. Once staff has confirmed that the two participants are a couple, they will be contacted to schedule an in-person meeting where they will complete a consent form and the baseline assessment.

Baseline Assessment. After couple confirmation, the couple will be scheduled for an in-person appointment. After consenting to participate in the study in-person (consent process described below), the 2 partners will be directed to complete a baseline assessment. This approximately 60-minute questionnaire will assess demographics, relationship characteristics, HIV knowledge and motivations, HIV risk and prevention behaviors, and other relevant psychosocial outcomes (e.g., substance use, mental health). The couple will then be given additional information about the structure of the intervention and scheduling options. The baseline assessment will occur 1 week prior to the first session of the 2GETHER intervention. Urethral/rectal STI testing will also occur at baseline.

Randomization. Dyads will be randomized to the 2GETHER intervention or attention-matched control using stratified block randomization, which involves performing simple randomization many times within blocks (e.g., ABBA, AABB, etc.), ensuring equal N in each condition while avoiding temporal imbalance. The eligibility screener will assess age and known HIV status. Blocks will be stratified to ensure equal numbers of couples assigned to each condition in which: (a) at least 1 member is HIV+; and (b) 1 member is aged 30+. Randomization will occur at completion of baseline survey. Baseline interviews will occur 1 week prior to 2GETHER/control session 1, and dyads will only be baselined if they are available for all sessions. Scheduling conflicts arise; 2 group cohorts are run simultaneously, so dyads that miss a group session can be scheduled for the same session in the other cohort.

2GETHER Intervention: The study intervention will take place over the course of 4 weeks (4 sessions total; approximately 1 session per week), beginning with 2 group sessions and ending with 2 individual couple sessions. During group sessions, 4-8 couples will work with 2 facilitators; in the couple's sessions, each individual couple will work with a single facilitator. Intervention content will be delivered via a combination of facilitated discussion, group and/or couple activities, worksheets, videos, and didactic material. Skills will be reinforced using interactive homework assignments between sessions, which will be reviewed at the beginning of the subsequent session. After each session, participants will complete a brief online evaluation to assess acceptability of the intervention content.

Session 1. The first group session (4 hours) will consist of four modules: 1) an orientation to the intervention, 2) characteristics of healthy relationships, 3) effective communication skills, and 4) reducing HIV risk in relationships. In the orientation module, couples will learn about the structure and purpose of the intervention, collaboratively develop a list of group rules with the facilitators (e.g., confidentiality, respect for others), and will complete ice-breaker activities to facilitate participants' comfort with the other group members. In the healthy relationships module, couples will learn how to identify healthy and unhealthy relationship patterns, discuss past experiences with healthy/unhealthy relationships, and then develop a list of pleasurable activities in which couples can engage in the Chicago area (e.g., free museum nights). Couples will identify one activity they will do in the next week. In the effective communication skills module, couples will learn about several effective and ineffective communication patterns, watch brief videos demonstrating these patterns, and briefly practice effective communication skills with their partners. Couples will be asked to practice using effective communication skills and identify instances in which they use ineffective communication with their partners before the next session. Finally, in the reducing HIV risk module, couples will learn about HIV risks in same-sex male relationships, sexual behaviors that pose different levels of HIV risk, different methods of HIV prevention including condom use, pre-exposure prophylaxis (PrEP), and post-exposure prophylaxis (PEP), and where one can be tested for HIV and obtain condoms and PrEP/PEP.

Session 2. The second group session (2 hours) will cover 1) coping skills, 2) problem-solving,3) social and community support, and 4) acceptance. In the coping skills modules, couples will learn the various types of strategies that can be used to cope with stress and will discuss which strategies are the most effective in various situations. In the problem-solving module, couples will learn a simple framework for addressing problems and stress in their relationship. In the social and community support module, couples will participants identify the social networks and communities that can serve as additional support for each individual and the couple. Finally, the acceptance module will teach couples who to identify stresses that can't be changed and will review strategies for accepting stressful situations without changing them in order to reduce their impact on the health of the couple.

Session 3. The first couples' session (1 hour) will consist of more in-depth discussion and practice of communication skills. Facilitators will elicit reasons why utilizing effective communication and minimizing ineffective communication are important for each couple, as well as ways in which using effective or ineffective communication has affected their relationship in the past. Couples will identify two areas of conflict or disagreement that can be targeted in a 30-minute skills practice. Each partner will take at least 1-2 turns communicating their concerns about the disagreement, listening to their partner communicate their concerns, and responding to their partner's concerns respectfully. The facilitator will provide each partner with feedback. Before the next session, couples will be asked to continue practicing effective communication on 1-2 additional topics identified in this session, to continue identifying and rectifying ineffective communication, and engage in another positive activity as a couple.

Session 4. The second couples' session (1.5 hours) will be focused on relationship sexual agreements. Couples will engage in a facilitated discussion about their perceived risk of HIV and identify their motivations for reducing HIV risk in their current relationship and/or with outside partners. Couples will learn about relationship agreements (i.e., agreements about whether or not it is permissible to have sex with partners outside of the relationships) and generate list of pros and cons about having outside partners and having relationship agreements in general. Couples who do not have a relationship agreement will, with the help of the facilitator, begin drafting an agreement that meets each partner's emotional, sexual, and health needs. Couples who have an existing agreement will identify whether their current relationship agreement meets these needs and determine whether and how to amend their relationship agreement. Couples will also learn about how relationship agreements may change over time, how to renegotiate agreements, how to communicate about a broken agreement, and how different agreement types impact HIV risk. Finally, the facilitator will review strategies for maintaining healthy relationships in the long-term, including discussing strategies the couples can use to handle lapses in their newly acquired healthy relationship skills.

Positive Affect Promotion Program (Control Condition):

The control condition will be a positive affect program developed by Co-I Dr. Moskowitz, that matches attention and the mixed group and individual format of 2GETHER. Developed based on Stress and Coping Theory and the Broaden-and-Build theory of positive emotion, this program aims to reduce distress and improve wellbeing by increasing attention to positive emotions and reducing impact of negative emotions. In this trial, Sessions 1 and 2 will be group sessions facilitated by two individuals and focused on didactic instruction of strategies for increasing positive affect in both individuals and couples. Analogous to 2GETHER, Sessions 3 and 4 will be individual couple sessions facilitated by one individual that focus on skills implementation in the dyad. Justification: The positive affect program has received high acceptability ratings and has been found to improve psychological distress in HIV+ MSM, but analyses find no effect on transmission risk behavior and we would not anticipate it would do so among HIV- MSM. This control condition is both ethical and appropriate for this RCT: it delivers beneficial skills but it does not address the primary mechanisms of change in 2GETHER (i.e., communication, sexual health negotiation skills). Exit interviews from our pilot trial indicate that this positive affect intervention would be beneficial to coupled YMSM but would not address 2GETHER's mechanisms of change: "I like the thought of learning to be more mindful, and I think that would be easier to do in a group setting, so we would enjoy the program. But I also feel that the new topics are less focused on communicating effectively as a couple, so I do not feel it would have had the same effect for me personally." Facilitators. Facilitators will hold a bachelor's degree at minimum and have direct experience working with young adults and/or MSM. Facilitators will receive project- and university-specific training and will be certified in HIV testing and counseling. Weekly supervision groups will review and discuss issues that arise during sessions. Using BA-level facilitators means 2GETHER will be easier to implement in the community.

Post-Session Evaluations. After each of the 4 intervention sessions (or single sessions in control condition), participants will complete brief online evaluations that assess feasibility and acceptability of the intervention, as well as provide ratings of the facilitators. These surveys will be programmed in REDCap software, and links to the evaluations will be emailed to participants after completing each session of the intervention.

Assessment Timepoints. Baseline assessment will occur in-person. Each individual will complete informed consent separately to ensure both are willing/able to participate. Intermediate follow-up assessments will be completed remotely online (to minimize burden) at 3-, 6-, and 9-months; 12-month follow-up will be completed in-person to facilitate collection of biological endpoints (STI testing). All assessments will last approximately 45-60 minutes will assess the same or analogous constructs.

Fidelity. The study will use 2 strategies to ensure fidelity to the intervention manual. First, an independent assessor will sit in on 20% of group sessions. Second, the study will audio-record all individual couple's sessions, and an independent assessor will review 20% of sessions for fidelity. Independent assessors will complete a checklist indicating whether or not each component of each intervention session was completed by facilitators.

ELIGIBILITY:
Inclusion Criteria:

* Both members of the couple assigned male at birth and currently identify as male
* Both members of the couples at least 18 years of age; at least one between the ages of 18-29 years
* Both members of the couple identify one another as primary partners
* Couple has had oral or anal sex with one another in the past 3 months
* At least one member of the couple reports condomless anal sex with a serodiscordant or unknown status partner during the past 3 months
* Both members of the couple read and speak English at 8th grade level or better
* Both members have Internet access
* Both members audio recording of intervention sessions

Exclusion Criteria:

* Severe intimate partner violence

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — participants required to be assigned male at birth and currently identify as male
Enrollment: 256 (Actual)
Dates: Start 2017-08-21 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Condomless anal sex | Baseline, 3-, 6-, 9-, 12-months
  change in number of condomless anal sex acts with serodiscordant or unknown status partners
Sexual Agreement Concordance | Baseline, 3-, 6-, 9-, 12-months
  change in concordance between each member of the dyad in the rules of their sexual agreement (monogamy or non-monogamy agreement)
Sexual Agreement Breaks | Baseline, 3-, 6-, 9-, 12-months
  occurrence of breaks in the rules of couples' sexual agreement (monogamy or non-monogamy agreement)
Occurrence of Sexually Transmitted Infections | Baseline, 12-months
  the incidence (number of new cases or diagnoses) of Chlamydia and Gonorrhea at 12 months

SECONDARY OUTCOMES:
HIV Testing | Baseline, 3-, 6-, 9-, 12-months
  frequency of HIV testing among HIV-negative or unknown status participants
Antiretroviral Medication Adherence | Baseline, 3-, 6-, 9-, 12-months
  change in ART medication adherence among HIV-positive participants

OTHER OUTCOMES:
Pre-Exposure Prophylaxis | Baseline, 3-, 6-, 9-, 12-months
  initiation of pre-exposure prophylaxis among HIV-negative or unknown status participants
Pre-Exposure Prophylaxis Adherence | Baseline, 3-, 6-, 9-, 12-months
  change in pre-exposure prophylaxis adherence among participants who have initiation pre-exposure prophylaxis
HIV Viral Load | Baseline, 12-months
  change in serum viral load among HIV-positive participants
Relationship Satisfaction | Baseline, 3-, 6-, 9-, 12-months
  change in relationship satisfaction
Relationship Communication | Baseline, 3-, 6-, 9-, 12-months
  change in use of effective and ineffective communication

CONTACTS AND LOCATIONS:
Overall Officials: Michael E Newcomb, Ph.D., Principal Investigator — Northwestern University; Jim Carey, MPH, Study Director — Northwestern University; Ricky Hill, Ph.D., Study Director — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sullivan PS, Salazar L, Buchbinder S, Sanchez TH. Estimating the proportion of HIV transmissions from main sex partners among men who have sex with men in five US cities. AIDS. 2009 Jun 1;23(9):1153-62. doi: 10.1097/QAD.0b013e32832baa34. PMID 19417579
- [Background] Greene GJ, Fisher KA, Kuper L, Andrews R, Mustanski B. "Is this normal? Is this not normal? There's no set example": Sexual Health Intervention Preferences of LGBT Youth in Romantic Relationships. Sex Res Social Policy. 2015 Mar;12(1):1-14. doi: 10.1007/s13178-014-0169-2. PMID 25678895
- [Background] Jiwatram-Negron T, El-Bassel N. Systematic review of couple-based HIV intervention and prevention studies: advantages, gaps, and future directions. AIDS Behav. 2014 Oct;18(10):1864-87. doi: 10.1007/s10461-014-0827-7. PMID 24980246
- [Background] Markman HJ, Rhoades GK. Relationship education research: current status and future directions. J Marital Fam Ther. 2012 Jan;38(1):169-200. doi: 10.1111/j.1752-0606.2011.00247.x. PMID 22283386
- [Background] Newcomb ME, Macapagal KR, Feinstein BA, Bettin E, Swann G, Whitton SW. Integrating HIV Prevention and Relationship Education for Young Same-Sex Male Couples: A Pilot Trial of the 2GETHER Intervention. AIDS Behav. 2017 Aug;21(8):2464-2478. doi: 10.1007/s10461-017-1674-0. PMID 28083833
- [Derived] Smith MS, Greenawalt I, Moskowitz JT, Addington EL, Mustanski B, Newcomb ME. Results of a positive affect intervention for male couples: Change over time and effects on mental health. J Consult Clin Psychol. 2025 Jul;93(7):511-525. doi: 10.1037/ccp0000963. PMID 40587318
- [Derived] Newcomb ME, Swann G, Addington EL, Macapagal K, Moskowitz JT, Sarno EL, Whitton SW, Mustanski B. Randomized controlled trial of a relationship education and HIV prevention program for young male couples: Biomedical and behavioral outcomes. Health Psychol. 2025 Mar;44(3):297-309. doi: 10.1037/hea0001448. PMID 39992776
- [Derived] Smith MS, Newcomb ME. Substance Use and Relationship Functioning Among Young Male Couples. Arch Sex Behav. 2023 Jul;52(5):2097-2110. doi: 10.1007/s10508-023-02627-1. Epub 2023 Jun 23. PMID 37351709
- [Derived] Newcomb ME, Sarno EL, Bettin E, Conway A, Carey J, Garcia C, Hill R, Jozsa K, Swann G, Addington EL, Ciolino JD, Macapagal K, Moskowitz JT, Mustanski B, Whitton SW. Protocol for an attention-matched randomized controlled trial of 2GETHER: a relationship education and HIV prevention program for young male couples. Trials. 2022 Jun 20;23(1):514. doi: 10.1186/s13063-022-06457-9. PMID 35725624